CLINICAL TRIAL: NCT05982418
Title: Improvement of Robotic-assisted Radical Prostatectomy (RARP) Outcomes Via Automatedly Segmented 3D Printed and Virtual Prostate Models: a Feasibility Study
Brief Title: Improvement of RARP Outcomes Via 3D Printed/Virtual Prostate Models
Acronym: RARP-3D
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Guy's and St Thomas' NHS Foundation Trust (Other)
Collaborators: King's College London (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 152847
Record Dates: First submitted 2023-07-20; First posted 2023-08-08 (Actual); Last update posted 2023-08-08 (Actual); Status verified 2022-12

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Intervention Model Description: A total of 108 patients will be recruited prospectively, i.e. 54 patients for intervention arm 1 (3D printed models), and 54 patients for intervention arm 2 (3D virtual models). An additional set of 54 patients will be obtained retrospectively.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 3D Printed Models (Experimental): This cohort will consist of 54 prospective cases whereby patient-specific 3D printed models will be available to the surgeon during RARP for manipulation.
  Interventions: Device: 3D Printed Models (3D printing facilities at GSTT)
- 3D Virtual Models (Experimental): This cohort will consist of 54 prospective cases whereby 3D virtual models will be available to the surgeon during RARP for manipulation using Innersight Labs platform.
  Interventions: Device: 3D Virtual Models (Innersight Labs)

INTERVENTIONS:
Device: 3D Printed Models (3D printing facilities at GSTT) — 3D patient-specific printed models are given to the surgeon before the start of RARP on a given patient. These 3D models are generated using automatic segmentation in MONAI followed by validation by a radiologist, and then post-processed for 3D printing.
  Arms: 3D Printed Models
Device: 3D Virtual Models (Innersight Labs) — 3D patient-specific virtual models loaded into Innersight Labs platform are given to the surgeon before the start of RARP on a given patient. These 3D models are generated using automatic segmentation in MONAI followed by validation by a radiologist, and then post-processed for 3D visualisation.
  Arms: 3D Virtual Models

SUMMARY:
Study the effect 3D printed or 3D virtual prostate models of a patient, when manipulated by surgeons during RARP, has on positive surgical margins and functional outcomes of patients. Our main hypothesis is that there is a reduction of positive resection margins and functional outcomes of patients undergoing RARP when surgeons are presented with 3D printed or 3D virtual patient-specific prostate models during surgery. Specifically, we hypothesize that the anatomical knowledge of surgeons that results from the manipulation of 3D printed/virtual models constructed from automated segmentations reduces positive resection margins and functional outcomes.

DETAILED DESCRIPTION:
This is a parallel group research feasibility study consisting of two intervention arms (3D printed and 3D virtual models) and a control group (standard practice). Intervention groups are prospective; control group is retrospective. Prospective patients, complying with the inclusion criteria, will randomly be allocated to only one intervention group.

Primary outcomes Study the effect of two-intervention arms (3D printed and virtual prostate models) have on the improvement of positive resection margins after RARP, validate the accuracy of automated methods when identifying masks of the prostate gland and, cancer lesions urethra, neurovascular bundles, and external sphincter, and validate the effectiveness of an automated deployment pipeline with the goal of setting groundwork in preparation for a randomise control trial in a subsequent study.

Secondary outcomes Study the effect of two-intervention arms have on functional outcomes, surgeons' and patients' perspectives on using 3D prostate models.

A total of 162 cases will be considered in this feasibility study stratified into 3 cohorts:

* Control group. The control group will consist of 54 retrospective case-matched dataset whereby mp-MRI, positive resection margins, and functional outcomes will be collected and used as a baseline. Automated segmentation of prostate gland and lesions will be done on mp-MRI.
* Intervention arm 1 - 3D printed models. This cohort will consist of 54 prospective cases whereby patient-specific 3D printed models will be available to the surgeon during RARP for manipulation.
* Intervention arm 2 - 3D virtual models. This cohort will consist of 54 prospective cases whereby 3D virtual models will be available to the surgeon during RARP for manipulation using Innersight Labs platform.

ELIGIBILITY:
Inclusion Criteria:

* Eligible for RARP after assessment of mp-MRI during multi-disciplinary team meetings at Guy's Hospital
* T2b-T3 prostate cancer patients
* Gleason's score>=3+4 .

Exclusion Criteria:

* prior treatment for prostate cancer
* patients with pre-existing urinary incontinence problems
* patients where mp-MRI scans are not possible
* patients participating in other studies investigating functional outcomes after surgery will be excluded. This is to avoid other studies influencing our secondary endpoints.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 162 (Estimated)
Dates: Start 2023-07-31 (Estimated); Primary Completion 2024-01-31 (Estimated); Study Completion 2024-01-31 (Estimated)

PRIMARY OUTCOMES:
Automated segmentation metrics | Assessed after mp-MRI of patient is available and before surgery (RARP). Reported at end of study (6 months).
  Automated segmentation metrics in relation to the accuracy of predicted masks of prostate gland and lesions
Patient recruitment rate | Assessed throughout the study for each patient. Reported at end of study (6 months).
  Patient recruitment rate will be captured throughout the study to measure effectiveness in preparation for a follow-up randomised control trial.
Percentage of cases that led to successful model deployment to the theatre | Assessed throughout the study for each patient. Reported at end of study (6 months).
  Percentage of cases that led to successful model deployment to the theatre will be captured throughout the study to measure effectiveness in preparation for a follow-up randomised control trial.
Positive resection margins | Duration of the study
  Assessed after surgery and after specimen analysis. Reported at end of study (6 months).

SECONDARY OUTCOMES:
Urinary incontinence leak outcomes | Assessed at 6 weeks and 3 months after surgery. Reported at end of study (6 months)
  These are captured via questionnaires (ICIQ-UI) answered by patients in relation to urinary leaks.
Urinary incontinence pad weights outcomes | Assessed at 6 weeks and 3 months after surgery. Reported at end of study (6 months)
  These are captured via questionnaires (EPROM) answered by patients in relation to urinary incontinence measured by pad weights.
Urinary incontinence quality of life outcomes | Assessed at 6 weeks and 3 months after surgery. Reported at end of study (6 months)
  These are captured via questionnaires (ICIQ-LUTS-QoL) answered by patients in relation to quality of life resulting from urinary incontinence.
Erectile dysfunction functional outcomes | Assessed at 6 weeks and 3 months after surgery. Reported at end of study (6 months)
  These are captured via questionnaires (IIEF, and erectile hardness score) answered by patients in relation to erectile dysfunction.
Surgeon's perspectives | Assessed only once after surgery and once surgeon has participated in both arms. Reported at end of study (6 months)
  Surgeon's perspectives on the use of patient-specific 3D printed and virtual prostate models during surgery will be captured after surgery
Patient's perspectives | Assessed after surgery and after first clinical follow-up at 6 weeks. Reported at end of study (6 months).
  Patient's perspectives on the use of their patient-specific 3D printed and virtual prostate model after surgery will be captured after surgery during clinic review
Accuracy metrics for the automated segmentation of other structures | Assessed after mp-MRI of patient is available and before surgery (RARP). Reported at end of study (6 months).
  Accuracy metrics of a model that will automatically identify neurovascular bundles, urethra, and external sphincter based on manually identified masks on mp-MRI
Surgical phase and action recognition | Assessed and reported at end of study (6 months).
  Surgical phase and action recognition accuracy metrics of RARP endoscopic videos to understand the actions done leading to the reported complications

IPD SHARING:
Plan to Share IPD: No